CLINICAL TRIAL: NCT03341195
Title: To Evaluate the Role of Mobile Phone SMS Messages and Automated Calls in Improving Vaccine Coverage Among Children in Pakistan
Brief Title: Mobile Phone SMS Messages and Automated Calls in Improving Vaccine Coverage Among Children in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Grand Challenges Canada (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr Abdul Momin Kazi, Senior Instructor Research, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4320-Ped_ERC-16
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Tuberculosis; Polio; Diphtheria; Pertussis; Tetanus; Haemophilus Influenzae Type b Infection; Hepatitis B; Pneumococcal Infection
Keywords: SMS; Automated calls; Routine immunization; mHealth
MeSH Terms: conditions — Tuberculosis; Poliomyelitis; Diphtheria; Whooping Cough; Tetanus; Haemophilus Infections; Hepatitis B; Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial, four intervention arm and one control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. One way SMS messages. (Active Comparator): Parents/caregiver will receive one way educational/reminder/proactive SMS messages related to routine immunization once a week till 20 weeks of age.
  Interventions: Behavioral: SMS messages and automated calls
- 2. Two Way SMS messages (Active Comparator): Parents/caregiver will receive two way (interactive) educational/reminder/proactive SMS messages related to routine immunization once a week till 20 weeks of age-parents will have the option to reply and receive more information related to immunization through text messages.
  Interventions: Behavioral: SMS messages and automated calls
- 3. One way automated calls. (Active Comparator): Parents/caregiver will receive one way educational/reminder/proactive automated phone call related to routine immunization once a week till 20 weeks of age.
  Interventions: Behavioral: SMS messages and automated calls
- 4.Two way interactive automated calls (Active Comparator): Parents/caregiver will receive two way (interactive) educational/reminder/proactive automated phone call related to routine immunization once a week till 20 weeks of age-parents will have the option to reply and receive more information related to immunization through phone call.
  Interventions: Behavioral: SMS messages and automated calls
- 5. Control Arm (No Intervention): One time counseling at the baseline survey.

INTERVENTIONS:
Behavioral: SMS messages and automated calls — The intervention consists of SMS and automated calls based messages
  Arms: 1. One way SMS messages.; 2. Two Way SMS messages; 3. One way automated calls.; 4.Two way interactive automated calls

SUMMARY:
Routine childhood immunization (RCI) in Pakistan is well below the recommended coverage of 90% with rates as low as 16% in certain regions (Pakistan DHS 2012-3). This has led to continued polio transmission, large measles outbreaks and thousands of deaths from vaccine-preventable diseases (Kazi.Bull WHO 2016). Mobile phone communication is widespread in developing countries and has proven a potential method of directly connecting pregnant women and mothers to health services (Kharbanda. Expert Review of Vaccine 2014). The investigators propose conducting a mixed methods proof of concept cluster randomized trial (CRT) to assess the effectiveness of different types of SMS messaging and automated calls to improve RCI and understand the perceptions and barriers that may affect SMS and automated call-based interventions at participants levels. the investigators will conduct the study at urban and rural sites in Pakistan. The investigators will examine an important public health question - do low cost, automated SMS, and automated messages improve RCI coverage in resource-constrained settings? Further, investigators will compare the effectiveness of reminder, educational and interactive text messages for improving RCI and will generate socio-cultural data regarding the impact of participants health beliefs that will be important for setting up the appropriate interventions in other LMICs.

DETAILED DESCRIPTION:
SMS text messages have shown to be effective for mobile health or mHealth having a considerable impact on disease prevention efforts in developing countries. Mobile phone and SMS texting provide an excellent solution to challenges like travel and complex intercultural contact. SMS based interventions have been quite effective in different programs, particularly in treatment adherence, smoke cessation, health care appointment attendance, antenatal care attendance and compliance with immunization. In addition adding incentives to SMS messages have shown a positive association, however, there is a cost implication for scaling up this model at a country level. Given the mobile phone access and acceptability in the LMIC, there is great potential for SMS based intervention to improve Immunization coverage in LMIC setup.

One major reservation for SMS based interventions is the level of literacy. However, there has been mixed input related to the preference of phones calls as compared to text messages in populations of low literacy and resource-constrained settings. Mobile phone text messages in local languages, pictorial messages and in combination with a phone call can further reduce this gap.

Most of the studies evaluating the impact of text messages on vaccination have been conducted in the United States with a major focus on flu vaccine among children and teenagers. The participants covered in these studies are from low income background at an academic medical center and is quite different from resource constraint settings of LMICs due to poor immunization registries and electronic records. There is limited data from LMICs set up on the role of SMS based interventions for improvement of RI coverage and conventional one-way reminder text messages were used by most of the studies as the intervention. Overall very few investigators compared reminders, educational and interactive SMS messages related to childhood vaccination uptake. Although some of the investigators have shown some behavior change for improvement in vaccination coverage, more rigorous application of health behavior change model needs to be applied to understand the impact of reminder, educational and interactive messages on behavior change related to improvement in RI coverage. Very few studies have compared the effect of educational, reminders and interactive messages in improving uptake and on-time routine immunization.

In this study the investigators would like to examine an important public health question - do low cost, automated SMS messages and calls improve RI coverage among participants in resource-constrained settings? In this study, we would like to compare the effectiveness of reminder, educational and interactive text messages and phone calls for improving RI uptake in Pakistani participants.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria includes being a child from the HDSS site, being less than 14 days of age with parent/guardian or at least one person in the household having a working mobile phone connection and parent/guardian providing consent to participate in the study.

Exclusion Criteria:

* The exclusion criteria includes a child from outside HDSS area or family plans to stay in the catchment area for less than 20 weeks

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3850 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will measure the number of children who got vaccinated for routine immunization scheduled at 6, 10 and 14 weeks of life | Vaccination status at 20th week of life of the particpants
  The final outcome of vaccine will be measured at 20 weeks of life, between control and intervention arm and between intervention arms

SECONDARY OUTCOMES:
The secondary outcome will measure the mean improvement in on-time vaccination for routine immunization scheduled at 6, 10 and 14 weeks of life | On-time vaccination for routine immunization scheduled at 6, 10 and 14 weeks of life
  The final outcome of on-time vaccination will be measured between control and intervention arm and between intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Abdul M Kazi, MBBS,MPH, Principal Investigator — The Aga Khan University, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Kazi AM, Ahsan N, Khan A, Jamal S, Kalimuddin H, Ghulamhussain N, Wajidali Z, Muqeet A, Zaidi F, Subzlani M, McKellin W, Ali A, Collet JP. Personalized Text Messages and Automated Calls for Improving Vaccine Coverage Among Children in Pakistan: Protocol for a Community-Based Cluster Randomized Clinical Trial. JMIR Res Protoc. 2019 May 30;8(5):e12851. doi: 10.2196/12851. PMID 31148544